CLINICAL TRIAL: NCT05440864
Title: Perioperative Therapy With Durvalumab Plus Tremelimumab for Patients With Resectable Hepatocellular Carcinoma (HCC) - A Phase II Trial (NEOTOMA)
Brief Title: Durvalumab and Tremelimumab in Resectable HCC
Acronym: (NEOTOMA)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Clinica Universidad de Navarra, Universidad de Navarra (Other); University of Milan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-5353
Record Dates: First submitted 2022-06-21; First posted 2022-07-01 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: hcc; resection; Durvalumab; Tremelimumab; neoadjuvant; adjuvant; phase II; perioperative; surgical; immunotherapy; hepatoma; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Intervention Model Description: This is a phase II, open label single arm, multicentre study of single dose Tremelimumab (T300) in combination with Durvalumab preoperatively in patients with upfront resectable HCC followed by adjuvant Durvalumab.
  This study will enroll 28 patients at three academic institutions in Canada and Europe. Patients will receive 1 dose Tremelimumab (300 mg) with Durvalumab (1500mg) at cycle 1 (4W) and 1 further cycle of Durvalumab (1500mg) pre surgical resection. Post-surgical resection patients will begin adjuvant Durvalumab (1500mg Q4W) to complete 13 cycles of treatment (or 11 post operatively) in total.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tremelimumab in combination with Durvalumab preoperatively, followed by adjuvant Durvalumab (Experimental): Patients will receive 1 dose Tremelimumab (300 mg) with Durvalumab (1500mg) at cycle 1 (4W) and 1 further cycle of Durvalumab (1500mg) pre surgical resection. Post-surgical resection patients will begin adjuvant Durvalumab (1500mg Q4W) to complete 13 cycles of treatment (or 11 post operatively) in total.
  Interventions: Drug: Tremelimumab

INTERVENTIONS:
Drug: Tremelimumab — Pre-operatively Tremelimumab will be administered first for 1 hour; the Durvalumab infusion (1hr) will start approximately 1 hour (maximum 2 hours) after the end of the Tremelimumab infusion. Post-operatively patients will receive Durvalumab Q4W to complete up to 12 months of treatment or a maximum of 11 cycles of adjuvant Durvalumab
  Other Names: Durvalumab

SUMMARY:
Hepatocellular Carcinoma (HCC) is the third most common cause of death from cancer world wide and the incidence is rising globally. Despite surgical resection in appropriate patients, many patients recur.

The results of the IMbrave150 study have established PD-L1 inhibition in combination with VEGF inhibition as a new standard of care highlighting the role of immune checkpoint inhibition in advanced HCC. In addition, the combination of Tremelimumab and Durvalumab has demonstrated efficacy in advanced HCC; the HIMALAYA trial has now completed accrual in treatment naïve patients with advanced HCC. Furthermore the earlier use of immune checkpoint inhibitors in this disease are being explored with adjuvant combination strategies, including the EMERALD-2 trial (NCT03847428). Neoadjuvant treatment in HCC allows for delivery of treatment pre surgery and may enhance pathological responses and improve outcomes. The delivery of combination CTLA-4 and PD-L1 inhibition has demonstrated efficacy in other tumour types in the neoadjuvant setting where the impact on the tumour microenvironment has also been evaluated. The safety and feasibility of Durvalumab and Tremelimumab in resectable HCC has yet to be established.

Hypotheses Pre-operative (pre-op) Durvalumab and Tremelimumab treatment is safe and feasible in pre surgical setting for upfront resectable HCC The combination of Durvalumab and Tremelimumab pre-op will result in changes in immune and molecular characteristics within the tumour microenvironment.

Overall Study Design This is a phase II, open-label multi-centre study to assess safety of Durvalumab and Tremelimumab treatment in pre-op setting for upfront resectable HCC, followed by adjuvant Durvalumab.

28 patients are expected to enrol at three sites. Patients will receive pre-op: 1 dose Tremelimumab (300mg) (T300) with Durvalumab (1500mg) at cycle 1 and 1 further cycle of Durvalumab (1500mg) only. Post-surgical resection, adjuvant therapy will consist of Durvalumab Q4W for up to a maximum of 12 months in total or 13 cycles of Durvalumab (11 cycles post op).

All participants will be treated until progressive disease or unacceptable toxicity or withdrawal of consent or another discontinuation criterion is met. All participants will be followed for survival until the end of study.

No dose reductions of Tremelimumab and Durvalumab will be allowed. Statistics The primary objective of this study is to assess safety of pre-op treatment with Durvalumab and Tremelimumab.

For safety, with the null proportion of patients who discontinue treatment due to AEs, imAEs or SAE is 30% versus the alternative proportion is 10% or less than 10%, a sample size of 28 provides 80% power to detect the proportion difference with a two-sided alpha level of 0.1.

The sample size estimate is based on the two-sided exact test for binomial proportion considering Binomial Enumeration method.

DETAILED DESCRIPTION:
INTRODUCTION This is a phase II, open label single arm, multicentre study of Tremelimumab in combination with Durvalumab (IMFINZI) in preoperative patients with resectable hepatocellular carcinoma (HCC) followed by adjuvant Durvalumab.

Disease background: HCC represents the third most common cause of cancer-related death and accounts for over 80% of primary liver cancers worldwide. Treatments are numerous and are selected based on tumour extent, patient comorbidities, and liver dysfunction. Surgical resection is recommended in patients with resectable tumours with otherwise well-compensated liver disease in the absence of clinically significant portal hypertension (hepatic vein to portal system gradient >10 mmHg or a platelet count ≤100,000/ml). Patients with macrovascular invasion, multifocal disease (within the same lobe), or large tumours that would require vascular resections and reconstructions are not typically considered for surgical resections according to the current clinical management guidelines. They are instead generally recommended to undergo systemic or locoregional therapies for palliation if they are not otherwise candidates for liver transplantation. In more favorable conditions of liver-confined disease and an absence of macrovascular invasion, still, many patients are deemed unresectable. Within this setting, strategies that can downstage tumors to allow resection to be performed, and help decrease the postoperative disease recurrence risk, are urgently needed. Moreover, when surgically resected, as many as 70% of the patients develop disease recurrence. Unfortunately, there are few clinical variables available that can aid in predicting postoperatively recurrence risk, many of which are only available on the pathology specimen after the liver resection has been performed, such as microvascular invasion or the presence of satellite lesions. A preoperative tumour biopsy, may identify biomarkers to immune checkpoint inhibitor response that can further help to refine treatment selection and potentially a subset of patients where neoadjuvant immune checkpoint inhibitor therapy use may be particularly beneficial. There is typically no discrepancy between the number of patients intended to receive liver resection and those who can undergo resection (i.e., no dropout while awaiting a liver resection). Consequently, given that the risk of tumour progression while awaiting surgical resection is low, the addition of neoadjuvant therapy during this wait is unlikely to lead to patients being unable to undergo their intended liver resection.

Study Rationale In advanced HCC combination immunotherapeutic strategies are rapidly becoming a new standard of care. The rationale for the use of immunotherapy in HCC is supported by the high expression of immunosuppressive cells, including PD-L1 expression, which is a poor prognostic factor. Therefore targeting immune checkpoints may improve outcomes, and several adjuvant trials are currently accruing patients.

Tremelimumab is a human IgG2 monoclonal antibody (mAb) directed against CTLA-4. The CTL-associated antigen 4 (CTLA-4) is an inhibitory receptor for B7, acting as an immune checkpoint resulting in a downregulation in T-cell activation through the competition with CD28 for B7 binding. Notably different to its IgG1 mAb counterparts, Tremelimumab may have less potential for antibody dependent cell mediated toxicity. Tremelimumab has previously been evaluated in hepatitis C-virus related HCC in a phase 2 trial .Twenty patients were included in the study, which reported a partial response rate of 17.6% and a disease control rate of 76.4%. Time to progression was 6.48 months (95% CI 3.95-9.14). In a phase 1/2 trial, evaluated the use of Tremelimumab in combination with ablation in patients with advanced HCC. Nineteen of the thirty-two patients enrolled were evaluable. Of these, five (26.3%, 95% CI 9.1-51.2%) achieved a partial response. In patients in whom a clinical benefit was observed, tumor biopsies at six weeks demonstrated an increase in CD8+ T cells. Six and 12-month tumor progression-free survival probabilities were 57.1% and 33.1%, respectively. The median OS was 12.3 months (95% CI 9.3-15.4 months). No dose-limiting toxicities were observed.

Durvalumab is a human immunoglobulin G1 kappa monoclonal antibody which blocks the interaction between the programmed cell death ligand 1 (PD-L1) (a member of the B7 family) with PD-1 (CD279). PD-L1 is expressed on several cells, including dendritic cells, macrophages, and many human cancer cells. PD-1 upregulation has been demonstrated on effector CD8+ T-cells in HCC. Moreover, both PD-1 and PD-L1 upregulation has been found to portend a poor prognosis in patients with HCC following surgical resection. In an interim analysis of a phase 1/2 trial of Durvalumab as monotherapy in HCC, out of forty patients, treatment-related adverse events occurred in 80.0% . Grade 3-4 treatment-related adverse events were reported in 20% of patients. Four patients achieved a partial response, and the objective response rate (complete response + partial response) was 10.3% (95% CI 2.9-24.2). Median OS was 13.2 months (95% CI 6.3-21.1). Following this, initial results of Study 22 a phase 1/2 randomized study were reported on Durvalumab and Tremelimumab in unresectable HCC (NCT02519348). In an updated analysis of Study-22 presented at the ASCO annual meeting longest survival in the advanced HCC population was reported with priming dose Tremelimumab 300mg x 1 dose (T300) in combination with Durvalumab 1500mg every four weeks. The overall response rate was 24% and median time to response 1.86 months. Median OS in this arm (18.7 months) was superior to single agent ICI and to low dose Tremelimumab in combination with Durvalumab. Eight patients or 10.8% stopped study due to treatment related adverse events. The HIMALAYA study, a randomized, multicenter phase 3 study of Durvalumab and Tremelimumab (300mg priming dose) as first-line therapy in unresectable HCC is closed to accrual.

Neoadjuvant therapy is commonly used in other solid-organ malignancies for three main reasons: downstage patients with advanced disease and to target micrometastatic disease, ensure patients are appropriately selected for curative treatment, and to evaluate tumour response to treatment before surgery. The role of neoadjuvant therapy in potentially resectable HCC is not clearly defined. Nonetheless, the aggressive biology of HCC, with high rates of tumour recurrence and de novo tumours after curative-intent resection, along with high immunosuppressive cell expression and CTLA-4 and PD-1 immune checkpoint upregulation, an investigation of the role of neoadjuvant immunotherapy in patients who present with resectable disease is warranted. Such treatment sequencing has demonstrated encouraging results in other lethal malignancies, such as non-small cell lung cancer. For example, evaluated the use of neoadjuvant PD-1 blockade (Nivolumab) in resectable (stage I, II, or IIIA) lung cancer (non-small-cell) in a pilot study. Nivolumab in the neoadjuvant setting had a side-effect profile that was acceptable and did not delay surgery. Complete surgical resection was obtained in 20 of the 21 tumors that were resected. Nine out of these twenty tumors (45%) demonstrated a major pathological response, which was correlated to the pre-treatment tumor mutational burden. Moreover, treatment with PD-1 blockade resulted in the expansion of mutation-associated, neoantigen-specific T-cell clones in peripheral blood.

Research hypothesis

* Pre-operative Durvalumab and Tremelimumab is safe in the pre surgical setting for upfront resectable HCC.
* Combination Durvalumab and Tremelimumab pre-operatively will result in changes in immune and molecular characteristics within the tumour microenvironment.

STUDY DESIGN This is a phase II, open label single arm, multicentre study of single dose Tremelimumab (T300) in combination with Durvalumab preoperatively in patients with upfront resectable HCC followed by adjuvant Durvalumab.

This study will enroll 28 patients at three academic institutions in Canada and Europe. Patients will receive 1 dose Tremelimumab (300 mg) with Durvalumab (1500mg) at cycle 1 (4W) and 1 further cycle of Durvalumab (1500mg) pre surgical resection. Post-surgical resection patients will begin adjuvant Durvalumab (1500mg Q4W) to complete 13 cycles of treatment (or 11 post operatively) in total.

Eligibility will be limited to patients with resectable HCC and preserved liver function. Prior systemic treatment for HCC will not be allowed although prior curative intent surgery or RFA is permitted.

All participants will be treated until progressive disease or unacceptable toxicity or withdrawal of consent or another discontinuation criterion is met. All participants will be followed for survival until the end of study.

No dose reductions of Durvalumab or Tremelimumab will be allowed. Dose modification and toxicity management for Durvalumab and Tremelimumab -related toxicity, including management of immune-mediated reactions, infusion-related reactions, and non-immune-mediated reactions will be provided in the Toxicity Management Guidelines (Appendix 1).

If the second cycle of Durvalumab is omitted due to toxicity, patients can resume adjuvant Durvalumab at the investigator's discretion and in accordance with protocol.

All patients enrolling will be required to undergo a pre-enrolment biopsy and for resected specimens will be required to provide consent to supply a sample of their tumor.

Scientific rationale for study design Rationale for primary endpoint The primary objective of this study is to assess the safety of Tremelimumab (T300) and Durvalumab pre-operatively in patients with resectable HCC followed by adjuvant Durvalumab (Q4W) for up to a maximum of 13 cycles or 11 post-operatively.Rationale for other secondary and exploratory endpoints The key secondary objectives are to evaluate feasibility, pathological response rates and overall response rates to pre-operative treatment.

Feasibility will be determined by the number of patients who had a delay in planned surgical resection (measured in days) due to TRAEs.

Major pathological response rates were recently demonstrated with the combination of CTLA-4 and PD-1 inhibition in resectable lung cancer. Furthermore, dynamic changes in immune correlates and microbiota composition were also documented.

Blood and tissue samples will be used to explore potential biomarkers in residual biological samples that may influence the progression of cancer and/or identify patients likely to have treatment benefit.

PD-L1 expression will be assessed and correlated with efficacy as a secondary objective. PD L1 is the target of Durvalumab, and it is hypothesized that its expression correlates with clinical efficacy.

Justification for dose Dose rationale for combination regimen of Durvalumab 1500mg Q4W plus Tremelimumab T300 The Durvalumab + Tremelimumab doses and regimen selected for this study are based on the goal of selecting an optimal combination dose of Durvalumab and Tremelimumab that would yield sustained target suppression (sPD-L1), demonstrate promising efficacy, and have an acceptable safety profile.

Rationale for 1 cycle of combination therapy with high dose Tremelimumab followed by Durvalumab monotherapy A summary of the existing PK and pharmacodynamic data has been utilized to guide the regimen selection for the combination of Durvalumab 1500 mg plus single dose of Tremelimumab 300 mg. Clinical Study Protocol Drug Substance Durvalumab (MEDI4736) and Tremelimumab Study Code D419CC00002 Version 1.0 Date 09 August 2017 39(219) Pharmacokinetics/pharmacodynamics data. The supporting data for this regimen are based on PK and pharmacodyamic data from regimens that used Tremelimumab doses of greater than 1 mg/kg from Study D4190C00006. An approximate dose-proportional increases in PK exposure (maximum plasma concentration and area under the plasma drug concentration-time curve from time 0 to Day 28 post-dose) was observed with increasing doses of Tremelimumab (1, 3, and 10 mg/kg). An exploratory pharmacodynamic analysis bioanalytically evaluated the effects of Tremelimumab on proliferating T-cells from NSCLC patients who received Tremelimumab (1, 3, or 10 mg/kg) and Durvalumab (15 or 20 mg/kg) combination treatment. Monotonic increases in pharmacodynamic activity with the combination (increased activation/ proliferation markers on CD4 and CD8 T-cells in periphery) were observed with increasing doses of Tremelimumab (1, 3, 10 mg/kg). The peak increase (%) from baseline of CD4+Ki67+ T-cells was observed 8 days post administration, and the peak level was significantly increased (p ≤ 0.05) as increasing dose of Tremelimumab in the range of 1 to 10 mg/kg. Study data also suggested that higher peak exposure (Cmax) of Tremelimumab is related to a higher maximum pharmacodynamic effect in the NSCLC patient population. Overall, the PK/pharmacodynamic data suggest that Tremelimumab of dose greater than 1 mg/kg with a higher peak exposure may be associated with a higher pharmacodynamic effect. Additionally, based on simulation data, the Cmax (78 µg/mL) post single dose administration of Tremelimumab 4 mg/kg is approximately 4-fold higher than the predicted Cmax (19 µg/mL) post the first dose of Tremelimumab 1 mg/kg, and is 3-fold higher than the predicted Cmax (25 µg/mL) post the fourth dose of Tremelimumab 1 mg/kg in a Q4W×4 doses setting.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients should fulfil the following criteria at time of study enrolment or when indicated:

1. Patient must be capable of providing written informed consent.
2. Age >18 years at time of study entry
3. Histologically proven resectable HCC (early and intermediate stage HCC)*
4. Must consent to provide biopsy sample prior to treatment
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
6. Childs Pugh score of 5 or 6
7. ALBI grade 1†
8. Patients with HBV infection, which is characterized by positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibodies (anti-HBcAb) with detectable HBV DNA (≥10 IU/ml or above the limit of detection per local lab standard), must be treated with antiviral therapy, as per institutional practice, to ensure adequate viral suppression (HBV DNA ≤2000 IU/mL) prior to study entry. Patients must remain on antiviral therapy for the study duration and for 6 months after the last dose of study medication. Patients who test positive for anti-hepatitis B core (HBc) with undetectable HBV DNA (<10 IU/ml or under limit of detection per local lab standard) do not require anti-viral therapy prior to study entry. These subjects will be tested at every cycle to monitor HBV DNA levels and initiate antiviral therapy if HBV DNA is detected (≥10 IU/ml or above the limit of detection per local lab standard). HBV DNA detectable subjects must initiate and remain on antiviral therapy for the study duration and for 6 months after the last dose of study medication.
9. Patients with HCV infection must have management of this disease per local institutional practice throughout the study. HCV diagnosis is characterized by the presence of detectable HCV ribonucleic acid (RNA) or anti-HCV antibody upon enrollment.
10. Evidence of post-menopausal status or negative serum pregnancy test for female pre-menopausal patients.
11. Female of childbearing potential and non-sterilized male partners of a female patient of childbearing potential must agree to use effective method of contraception from the time of screening throughout the total duration of the drug treatment and 6 months after the last dose of study treatment. (See exclusion #22 for definition of effective method of contraception).
12. Adequate normal organ and marrow function as defined below within screening period:

    * Haemoglobin ≥9.0 g/dL
    * Absolute neutrophil count (ANC ≥1.0 × 109 /L)
    * Platelet count ≥65 × 109/L
    * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). <<This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal
    * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

    Males:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) / 72 x serum creatinine (mg/dL)

    Females:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 / 72 x serum creatinine (mg/dL)

    - Albumin ≥2.8g/dl

    - International normalized ratio ≤1. (for patients receiving Warfarin, please consult with the study physician)
13. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
14. Body weight > 30kg

Exclusion Criteria:

* 1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.

  2. Any prior therapy for HCC - except liver resection or ablation on one occasion only which was given with curative intent and that occurred at least two years prior to study enrolment.

  3. Evidence of distant metastasis co-existing malignant disease or macrovascular invasion on baseline imaging.

  4. History of hepatic encephalopathy within 12 months prior to enrolment or requirement for medications to prevent or control encephalopathy (no lactulose, rifaximin, etc, if used for purposes of hepatic encephalopathy).

  5. Evidence of portal vein thrombosis, visible on baseline/eligibility imaging, and patients with Vp1, Vp2, Vp3 and Vp4.

  6. Clinically meaningful ascites, defined as ascites requiring non-pharmacologic intervention (eg, paracentesis) to maintain symptomatic control, within 6 months prior to the first dose of study treatment.

  (a) Patients with ascites who have required pharmacologic intervention (eg, diuretics) and who have been on stable doses of diuretics for ascites for ≥2 months before enrolment are eligible.

  7. Any history of nephrotic or nephritic syndrome. 8. Evidence of symptomatic congestive heart failure (New York Heart Association II to IV) or symptomatic or poorly controlled cardiac arrhythmia.

  9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [except for diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [e.g., granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, and uveitis]). The following are exceptions to this criterion:

  (a) Patients with vitiligo or alopecia (b) Patients with hypothyroidism (e.g., following Hashimoto syndrome), stable on hormone replacement (c) Any chronic skin condition that does not require systemic therapy (d) Patients without active disease in the last 5 years may be included but only after consultation with the Study Physician (e) Patients with celiac disease controlled by diet alone 10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active interstitial lung disease (ILD), serious chronic GI conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase the risk of incurring AEs or compromise the ability of the patient to give written informed consent.

  11. History of another primary malignancy except for the following:
  1. Prostate cancer of pathologic stage less than or equal to T2cN0M0 determined from a prior prostatectomy without biochemical recurrence and who, in the opinion of the Investigator, are not deemed to require active intervention, or patients with incidental histologic findings of prostate cancer that has not been treated prior to the study and who do not require specific therapy for prostate cancer beyond the surgery described in the Clinical Study Protocol and also are considered to be at low risk for recurrence per the Investigator
  2. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study treatment and of low potential risk for recurrence
  3. Adequately treated non-melanoma skin cancer or lentigo malignant without evidence of disease
  4. Adequately treated carcinoma in situ without evidence of disease 12. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.

     13. Active infection, including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice) or human immunodeficiency virus (HIV; positive for HIV 1/2 antibodies).

     14. Active co-infection with both HBV and HCV, or co-infected with HBV and hepatitis D virus.

     15. Known allergy or hypersensitivity to any of the study treatments or any of the study treatment excipients.

     16. Major surgery (as defined by the Investigator) within 28 days prior to enrolment, or central venous access device placement within 7 days prior to enrolment (biopsy from any type of surgery within 28 days is not an exclusion criteria, nor are procedures to treat varices).

     17. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart) 18. History of active primary immunodeficiency 19. History of allogeneic organ transplantation or those who are on a waiting list for liver transplantation.

     20. Receipt of live attenuated vaccine within 30 days prior to the first dose of study treatment. Note: Patients, if enrolled, should not receive live vaccine while receiving study treatment and up to 90 days after the last dose of study treatment.

     21. Current or prior use of immunosuppressive medication within 14 days before the first dose of study treatment. The following are exceptions to this criterion:

  (a) Intranasal, inhalational, topical steroids, or local steroid injections (e.g., intra-articular injection) (b) Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent (c) Steroids as pre-medication for hypersensitivity reactions (e.g., CT-scan premedication) 22. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 6 months after the last dose of study treatment. Not engaging in sexual activity, per the patient's preferred and usual lifestyle, for the total duration of the treatment and 6 months after the last dose of study treatment is an acceptable practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of greater than grade 3 adverse events (AEs) or immune related adverse events that leads to treatment cessation | 4 years
  Null proportion of patients who discontinue treatment due to AEs, imAEs or SAE is 30% versus the alternative proportion is 10% or less than 10%, a sample size of 28 provides 80% power to detect the proportion difference with a two-sided alpha level of 0.1.

SECONDARY OUTCOMES:
Number of patients who experience a surgical delay due to treatment related adverse events (TRAEs) | 4 years
Overall response rate (ORR) | 2 year
  According to RECIST v1.1 and mRECIST Objective response rate (ORR)
Pathological response rate | 2 year
  Percentage of Viable tumour remaining
Rates of R0 resection | 2 year
  Number of resections with negative margins

OTHER OUTCOMES:
Recurrence free survival | 4 years
  Recurrence free survival using RECIST 1.1
Overall survival | 4 years
  Overall survival
Changes in immune markers in tissue collected | 4 years
  To evaluate changes in immune markers in tissue collected both - pre-treatment and post-treatment with Durvalumab and Tremelimumab
PD-L1 expression | 4 years
  To establish PD-L1 expression using IHC pre and post Durvalumab and Tremelimumab
Durvalumab and Tremelimumab and blood biomarkers expression | 4 years
  To explore associations between exposure to Durvalumab and Tremelimumab and blood biomarkers.
Taxonomic profiling of gut microbiome | 4 years
  To evaluate taxonomic profiling of gut microbiome pre and post Durvalumab and Tremelimumab treatment and on adjuvant Durvalumab

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Sapisochin, MD, Study Chair — Univeristy Health Network; Grainne O'Kane, MD, Study Chair — Univeristy Health Network; Jennifer Knox, MD, Principal Investigator — Univeristy Health Network; Bruno Sangro, MD, Principal Investigator — Clinica Universidad de Navarra; Vincenzo Mazaferro, MD, Principal Investigator — University of Milan
Locations (3):
- University Health Network, Toronto, Ontario, Canada
- University of Milan, Milan, Italy
- Clinica Universidad De Navarra, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang JD, Hainaut P, Gores GJ, Amadou A, Plymoth A, Roberts LR. A global view of hepatocellular carcinoma: trends, risk, prevention and management. Nat Rev Gastroenterol Hepatol. 2019 Oct;16(10):589-604. doi: 10.1038/s41575-019-0186-y. Epub 2019 Aug 22. PMID 31439937
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Background] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Background] Pinato DJ, Fessas P, Sapisochin G, Marron TU. Perspectives on the Neoadjuvant Use of Immunotherapy in Hepatocellular Carcinoma. Hepatology. 2021 Jul;74(1):483-490. doi: 10.1002/hep.31697. Epub 2021 Jun 28. No abstract available. PMID 33369758
- [Background] Tabrizian P, Jibara G, Shrager B, Schwartz M, Roayaie S. Recurrence of hepatocellular cancer after resection: patterns, treatments, and prognosis. Ann Surg. 2015 May;261(5):947-55. doi: 10.1097/SLA.0000000000000710. PMID 25010665
- [Background] Golse N, Duarte P, Fontana A, Bundchen C, Karam V, Allard MA, Pittau G, Ciacio O, Duclos-Vallee JC, Sa Cunha A, Castaing D, Cherqui D, Adam R, Samuel D, Vibert E. Comparative analysis of outcomes after liver resection and liver transplantation for early stages hepatocellular carcinoma in HIV-infected patients. An intention-to-treat analysis. HPB (Oxford). 2020 Jun;22(6):900-910. doi: 10.1016/j.hpb.2019.10.014. Epub 2019 Nov 14. PMID 31734238
- [Background] Breous E, Thimme R. Potential of immunotherapy for hepatocellular carcinoma. J Hepatol. 2011 Apr;54(4):830-4. doi: 10.1016/j.jhep.2010.10.013. Epub 2010 Nov 9. PMID 21145836
- [Background] Greten TF, Sangro B. Targets for immunotherapy of liver cancer. J Hepatol. 2017 Sep 18:S0168-8278(17)32287-0. doi: 10.1016/j.jhep.2017.09.007. Online ahead of print. PMID 28923358
- [Background] Abou-Alfa GK CS, Furuse J, Galle PR, Kelley RK, Qin S, et al. . A randomized, multicenter phase 3 study of durvalumab (D) and tremelimumab (T) as first-line treatment in patients with unresectable hepatocellular carcinoma (HCC): HIMALAYA study. . J Clin Oncol 2018;36(15_suppl):TPS4144-TP4144. 2018.
- [Background] Gao Q, Wang XY, Qiu SJ, Yamato I, Sho M, Nakajima Y, Zhou J, Li BZ, Shi YH, Xiao YS, Xu Y, Fan J. Overexpression of PD-L1 significantly associates with tumor aggressiveness and postoperative recurrence in human hepatocellular carcinoma. Clin Cancer Res. 2009 Feb 1;15(3):971-9. doi: 10.1158/1078-0432.CCR-08-1608. PMID 19188168
- [Background] Arce Vargas F, Furness AJS, Litchfield K, Joshi K, Rosenthal R, Ghorani E, Solomon I, Lesko MH, Ruef N, Roddie C, Henry JY, Spain L, Ben Aissa A, Georgiou A, Wong YNS, Smith M, Strauss D, Hayes A, Nicol D, O'Brien T, Martensson L, Ljungars A, Teige I, Frendeus B; TRACERx Melanoma; TRACERx Renal; TRACERx Lung consortia; Pule M, Marafioti T, Gore M, Larkin J, Turajlic S, Swanton C, Peggs KS, Quezada SA. Fc Effector Function Contributes to the Activity of Human Anti-CTLA-4 Antibodies. Cancer Cell. 2018 Apr 9;33(4):649-663.e4. doi: 10.1016/j.ccell.2018.02.010. Epub 2018 Mar 22. PMID 29576375
- [Background] Sangro B, Gomez-Martin C, de la Mata M, Inarrairaegui M, Garralda E, Barrera P, Riezu-Boj JI, Larrea E, Alfaro C, Sarobe P, Lasarte JJ, Perez-Gracia JL, Melero I, Prieto J. A clinical trial of CTLA-4 blockade with tremelimumab in patients with hepatocellular carcinoma and chronic hepatitis C. J Hepatol. 2013 Jul;59(1):81-8. doi: 10.1016/j.jhep.2013.02.022. Epub 2013 Mar 4. PMID 23466307
- [Background] Duffy AG, Ulahannan SV, Makorova-Rusher O, Rahma O, Wedemeyer H, Pratt D, Davis JL, Hughes MS, Heller T, ElGindi M, Uppala A, Korangy F, Kleiner DE, Figg WD, Venzon D, Steinberg SM, Venkatesan AM, Krishnasamy V, Abi-Jaoudeh N, Levy E, Wood BJ, Greten TF. Tremelimumab in combination with ablation in patients with advanced hepatocellular carcinoma. J Hepatol. 2017 Mar;66(3):545-551. doi: 10.1016/j.jhep.2016.10.029. Epub 2016 Nov 2. PMID 27816492
- [Background] Wainberg ZA SN, Jaeger D, Lee K-H, Marshall J, Antonia SJ, et al. . Safety and clinical activity of durvalumab monotherapy in patients with hepatocellular carcinoma (HCC). . J Clin Oncol 2017;35(15_suppl):4071. 2017.
- [Background] Kelley RK SB, Harris WP, Ikeda M, Okusaka T, Kang YK, Qin S, Tai WM, Lim HY, Yau T, Yong WP. . Efficacy, tolerability, and biologic activity of a novel regimen of tremelimumab (T) in combination with durvalumab (D) for patients (pts) with advanced hepatocellular carcinoma (aHCC).
- [Background] Qin A, Coffey DG, Warren EH, Ramnath N. Mechanisms of immune evasion and current status of checkpoint inhibitors in non-small cell lung cancer. Cancer Med. 2016 Sep;5(9):2567-78. doi: 10.1002/cam4.819. Epub 2016 Jul 15. PMID 27416962
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Zhang C, Wu S, Xue X, Li M, Qin X, Li W, Han W, Zhang Y. Anti-tumor immunotherapy by blockade of the PD-1/PD-L1 pathway with recombinant human PD-1-IgV. Cytotherapy. 2008;10(7):711-9. doi: 10.1080/14653240802320237. PMID 18841514
- [Background] Rizvi NA, Mazieres J, Planchard D, Stinchcombe TE, Dy GK, Antonia SJ, Horn L, Lena H, Minenza E, Mennecier B, Otterson GA, Campos LT, Gandara DR, Levy BP, Nair SG, Zalcman G, Wolf J, Souquet PJ, Baldini E, Cappuzzo F, Chouaid C, Dowlati A, Sanborn R, Lopez-Chavez A, Grohe C, Huber RM, Harbison CT, Baudelet C, Lestini BJ, Ramalingam SS. Activity and safety of nivolumab, an anti-PD-1 immune checkpoint inhibitor, for patients with advanced, refractory squamous non-small-cell lung cancer (CheckMate 063): a phase 2, single-arm trial. Lancet Oncol. 2015 Mar;16(3):257-65. doi: 10.1016/S1470-2045(15)70054-9. Epub 2015 Feb 20. PMID 25704439
- [Background] Pardee AD, Butterfield LH. Immunotherapy of hepatocellular carcinoma: Unique challenges and clinical opportunities. Oncoimmunology. 2012 Jan 1;1(1):48-55. doi: 10.4161/onci.1.1.18344. PMID 22720211
- [Background] Antonia SJ BJ, Khleif S, et al. . Phase 1/2 study of the safety and clinical activity of durvalumab in patients with non-small cell lung cancer (NSCLC) [abstract no. 1216PD]. . Ann Oncol 2016;27(Suppl 6) doi:101093/annonc/mdw38316. 2016.
- [Background] Lee MS, Ryoo BY, Hsu CH, Numata K, Stein S, Verret W, Hack SP, Spahn J, Liu B, Abdullah H, Wang Y, He AR, Lee KH; GO30140 investigators. Atezolizumab with or without bevacizumab in unresectable hepatocellular carcinoma (GO30140): an open-label, multicentre, phase 1b study. Lancet Oncol. 2020 Jun;21(6):808-820. doi: 10.1016/S1470-2045(20)30156-X. PMID 32502443